CLINICAL TRIAL: NCT02369718
Title: Consequences of Aging and Dirtying of Microphones on the Performances of Cochlear Implants. Influence of Signal Coding
Brief Title: Cochlear Implants : Influence of Microphone Aging and Dirtying
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014.873
Record Dates: First submitted 2015-01-22; First posted 2015-02-24 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Hard of Hearing
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Implanted subjects (Experimental): Listening to 12 Fournier's lists of words
  Interventions: Other: Listening to 12 Fournier's lists of words
- Normal hearing subjects (Active Comparator): Listening to 48 Fournier's lists of words
  Interventions: Other: Listening to 48 Fournier's lists of words

INTERVENTIONS:
Other: Listening to 12 Fournier's lists of words — Patients will listen to words from Fournier's lists of words in presence of noise presented at different Signal to Noise Ratio (SNR). 6 disyllable words Fournier's lists are presented to the implantees: SNRs ranged from 0 to 15 decibels (dBs) (0; 3; 6; 9; 12; 15) ; the subjects repeat orally the words. Then microphone is cleaned and, again, 6 Fournier's lists are presented.
  Arms: Implanted subjects
Other: Listening to 48 Fournier's lists of words — 48 disyllable Fournier's lists of words are presented to the subjects (6 SNR*2 coding strategies*4 dirtying levels) and the subjects repeat orally the words. Dirtying levels will be simulated by sounds effects.
  Arms: Normal hearing subjects

SUMMARY:
Cochlear implant microphones are subject to aging and dirtying. The evolution may affect their efficiency. Several signal coding strategies are used in cochlear implants and their behaviour may be more or less affected by the aging process. In this work the investigators wish to assess this phenomenon.

ELIGIBILITY:
Inclusion Criteria:

* French speaking persons (French native speakers; studies made in French)
* Ear, Nose and Throat (ENT) tests and check up for normal hearing listeners were normal (Hearing loss below 20 dBs for all frequencies situated in the 250-8000 Hz range)
* Not mentally retarded

Exclusion Criteria:

* Persons with tinnitus or headache
* Anxious people (taking psychiatric drugs)
* Mental alteration or mental retard
* Deafened persons or taking an ENT treatment (normal hearing listeners)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2014-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Percentage of correct syllable recognition | At day 1
  French "spondee lists"

CONTACTS AND LOCATIONS:
Locations (1):
- Pavillon ORL (U) - Hôpital Edouard Herriot, Lyon, France

REFERENCES:
- [Background] P.A. Cucis, C. Berger-Vachon, E. Truy, H. Thai Van, F. Millioz, S. Gallego; "Cochlear Implants : Influence of the Coding Strategy on Syllable Recognition in Noise" AMSE JOURNALS-AMSE IFRATH Publication -2016: Modelling C; vol. 77; no 2; pp 84-97; 2016.
- [Background] P.A. Cucis, E. Veuillet, E. Truy, H. Thai Van, F. Millioz, S. Gallego; "Coding Strategy Robustness related to Microphone Integrityin Cochlear Implantsusing the Recognition of Syllables in a Noisy Environment"; AMSE JOURNALS-2016-Series: Advances B; vol. 59; no 1; pp 15-30; 2016.
- [Background] P.A. Cucis, E. Veuillet, E. Truy, H. Thai Van, F. Seldran, S. Gallego; "Effect of Microphone Cleaning on Syllable Recognition Performed by Cochlear Implant Users using the CIS and NofM Coding Strategies"; AMSE JOURNALS-2016-Series, Advances B; vol. 59; no 1; pp 31-45; 2016.
- [Background] P.A. Cucis, C. Berger-Vachon, E. Truy, H. Thai Van, F. Seldran, S. Gallego ; " Apport du nettoyage du microphone sur la reconnaissance de syllabes par des sujets implantés cochléaires selon les stratégies de codage CIS et N of M" ; Les Cahiers de l'Audition ; vol 29 ; no 5 ; pp 18-23 ; 2016.
- [Background] P.A. Cucis, C. Berger-Vachon, E. Truy, H. Thai Van, F. Millioz, S. Gallego " Influence de la stratégie de codage de l'implant cochléaire sur la reconnaissance de syllabes en milieu bruité en fonction de l'encrassement du microphone " Les Cahiers de l'Audition, vol 29, no 5, pp 12- 17, 2016.
- [Background] P.A. Cucis, C. Berger-Vachon, E. Truy, H. Thai Van, F. Millioz, S. Gallego; " Influence de la stratégie de codage de l'implant cochléaire sur la reconnaissance de syllabes en milieu bruité " Congrès Handicap 2016, IFRATH, Paris, 2016.